CLINICAL TRIAL: NCT07368244
Title: Turkish Translation and Content Validity of the Nottwil Environmental Factors Inventory (NEFI) in Persons With Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, Ass. Prof., Istanbul Medeniyet University
Other Study IDs: SCI NEFI-SF
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: InSCI; Nottwil Environmental Factors Inventory; NEFI; Turkish; cultural adaptation; content validity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational methodology study will produce a Turkish version of the Nottwil Environmental Factors Inventory (NEFI-TR) within one month using a standardized translation and cultural adaptation process. Content validity will be assessed using an expert panel (and, if applicable, cognitive debriefing with adults with spinal cord injury) to ensure relevance, clarity, and comprehensibility of each item in the Turkish context.

DETAILED DESCRIPTION:
Translation/adaptation: (1) two independent forward translations into Turkish; (2) reconciliation and harmonization by a multidisciplinary committee; (3) back-translation by independent translators; (4) expert committee review for semantic, idiomatic, experiential, and conceptual equivalence; (5) pre-test/cognitive debriefing (if planned) and final revisions; (6) proofreading and finalization of NEFI-TR and documentation of all decisions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>=16 years) with a diagnosis/history of spinal cord injury (traumatic or non-traumatic)
* Living in Turkey
* Able to read/understand Turkish and provide informed consent
* Clinically stable to complete questionnaires

Exclusion Criteria:

* Fully recovered from SCI / no longer living with SCI-related functional consequences (as defined by your protocol)
* Severe cognitive/communication limitations preventing valid completion
* Any condition judged by investigators to preclude participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (≥16 years) living in Turkey with a history of spinal cord injury (traumatic or non-traumatic) who can read and understand Turkish and provide informed consent. Participants will be recruited from rehabilitation/SCI outpatient settings and/or patient networks to complete the Turkish NEFI (NEFI-TR) pretest as part of the translation and content validity process. Individuals coded as fully recovered from SCI (i.e., no ongoing SCI-related limitations) will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Item Content Validity Index (I-CVI) | 1 month
  Item Content Validity Index (I-CVI) for NEFI-TR, derived from expert ratings of item relevance on a 4-point scale.
Scale Content Validity Index (S-CVI/Ave) | 1 month
  Scale Content Validity Index (S-CVI/Ave) for NEFI-TR, derived from expert ratings of item relevance on a 4-point scale.

SECONDARY OUTCOMES:
Qualitative feedback on clarity/comprehensibility | 1 month
  Qualitative feedback on clarity/comprehensibility; proportion of items requiring modification; (if cognitive debriefing) participant-rated clarity and acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Goztepe Prof Dr Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study is limited to questionnaire translation and content validity assessment and will use minimal, non-interventional data. Only aggregate, de-identified results (e.g., item-level content validity indices and summary statistics) will be reported.

REFERENCES:
- [Background] Yang Y, Gong Z, Reinhardt JD, Xu G, Xu Z, Li J. Environmental barriers and participation restrictions in community-dwelling individuals with spinal cord injury in Jiangsu and Sichuan Provinces of China: Results from a cross-sectional survey. J Spinal Cord Med. 2023 Mar;46(2):277-290. doi: 10.1080/10790268.2021.1935094. Epub 2021 Jun 17. PMID 34139132
- [Background] Ballert CS, Post MW, Brinkhof MW, Reinhardt JD; SwiSCI Study Group. Psychometric properties of the Nottwil Environmental Factors Inventory Short Form. Arch Phys Med Rehabil. 2015 Feb;96(2):233-40. doi: 10.1016/j.apmr.2014.09.004. Epub 2014 Sep 28. PMID 25264112
- [Background] Juvalta S, Post MW, Charlifue S, Noreau L, Whiteneck G, Dumont FS, Reinhardt JD. Development and cognitive testing of the Nottwil Environmental Factors Inventory in Canada, Switzerland and the USA. J Rehabil Med. 2015 Aug 18;47(7):618-25. doi: 10.2340/16501977-1982. PMID 26122005